CLINICAL TRIAL: NCT03576001
Title: Effect of a Multimodality Intervention to Improve Function and Metabolism in Spinal Cord Injury
Brief Title: Multimodality Intervention for Function and Metabolism in SCI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Spaulding Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Shalendar Bhasin, MD, Professor, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018P001431; R01HD093724-01 (NIH)
Record Dates: First submitted 2018-06-22; First posted 2018-07-03 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries | interventions — testosterone undecanoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Multi-modality intervention group (Experimental): Hybrid exercise (functional electrical stimulation - leg cycling, FES LC plus arm ergometry) plus Testosterone undecanoate
  Interventions: Drug: Testosterone Undecanoate; Behavioral: hybrid exercise
- Placebo group (Placebo Comparator): Hybrid exercise plus placebo medication
  Interventions: Behavioral: hybrid exercise

INTERVENTIONS:
Drug: Testosterone Undecanoate — administered through injections by study staff
  Arms: Multi-modality intervention group
Behavioral: hybrid exercise — hybrid exercise: functional electrical stimulation of lower extremity with leg cycling (FES-LC) and arm ergometry, supervised for two weeks and then home-based

SUMMARY:
The proposed phase 2 trial a randomized, placebo-controlled, parallel group trial in persons with cervical or thoracic SCI, AIS grade A, B, C, or D, 6 months or later after injury. The trial will test the hypothesis that a Home-Based Multimodality Functional Recovery and Metabolic Health Enhancement Program that addresses multiple pathophysiologic factors in SCI and includes functional electrical stimulation during leg cycling (FES-LC) plus arm ergometry and an androgen will be more efficacious than functional electrical stimulation during leg cycling (FES-LC) plus arm ergometry plus placebo in improving aerobic capacity, function, metabolism, bone health, and wellbeing.

DETAILED DESCRIPTION:
Study Description: The proposed phase 2 trial a randomized, placebo-controlled, parallel group trial in persons with cervical or thoracic SCI, AIS grade A, B, C, or D, 6 months or later after injury. The trial will test the hypothesis that a Home-Based Multimodality Functional Recovery and Metabolic Health Enhancement Program that addresses multiple pathophysiologic factors in SCI and includes functional electrical stimulation during leg cycling (FES-LC) plus arm ergometry and an androgen will be more efficacious than functional electrical stimulation during leg cycling (FES-LC) plus arm ergometry plus placebo in improving aerobic capacity, function, metabolism, bone health, and wellbeing.

Objectives:

Primary Objective:

• To determine whether the multimodality intervention is more efficacious in improving peak aerobic capacity, and muscle mass and strength than placebo plus functional electrical stimulation during leg cycling (FES-LC) plus arm ergometry alone.

Secondary Objectives:

* To determine whether the multimodality intervention is more efficacious than placebo plus functional electrical stimulation during leg cycling (FES-LC) plus arm ergometry in improving metabolic health, as reflected in fasting glucose, hemoglobin A1C, insulin sensitivity, fat mass and distribution, plasma lipids, and inflammation markers.
* To determine whether the multimodality intervention is more efficacious than placebo plus functional electrical stimulation during leg cycling (FES-LC) plus arm ergometry in improving volumetric and areal bone density, bone microarchitecture, and bone strength.

To determine the efficacy of the multimodality intervention in improving self-reported physical function (using SCI-FI AT and wellbeing (mood, anxiety, pain, loneliness and life satisfaction)

• To assess safety by structured monitoring of adverse events, and determining the proportion of participants experiencing injury, erythrocytosis, or other androgen-related or exercise-related adverse events.

Endpoints: Primary Endpoint:

Our primary outcome is peak aerobic capacity because it is an excellent marker of overall health, physical function, and mortality. Aerobic capacity is closely related to metabolic health, insulin sensitivity and cardiovascular outcomes. It can be measured accurately in SCI patients and would be expected to improve with the proposed interventions.

Secondary endpoints. Whole body skeletal muscle and fat mass and intraabdominal fat will be assessed by magnetic resonance imaging (MRI), using the Dixon method for separation of water/ fat signals. Body composition will also be measured by DEXA.

Maximal voluntary strength and muscle fatigability in the upper extremity will be assessed using the 1-repetition maximum in chest press.

Total, trabecular and cortical volumetric bone density; trabecular and cortical microarchitecture, both measured using high resolution peripheral quantitative computed tomography (HR-pQCT) at the ultradistal tibia, proximal tibia, and ultradistal radius.

Estimated bone strength of the ultradistal tibia and radius, assessed using microfinite element analysis of the HR-pQCT data.

Areal bone mineral density of the hip and lumbar spine using dual-energy X-ray absorptiometry (DEXA). (aBMD will be measured because DEXA is a clinically used and accepted measure of bone density, and aBMD is predictive of fracture risk.) Serum bone turnover markers, including markers of bone formation (osteocalcin, bone specific alkaline phosphatase (BSAP), (PINP) and bone resorption (CTX).

Spinal Cord Injury - Functional Index (SCI-FI) will be used to assess self-reported function and mobility. SCI-FI is specific for persons with SCI that assesses functional capacity in basic mobility, ambulation, self-care, and fine motor function, and wheelchair ambulation.

Measures of Metabolism: Fasting glucose, A1C; insulin sensitivity using HOMA-IR; IL-6 and hsCRP as inflammation markers; and plasma lipids, apolipoproteins B, C and A, and lipoprotein particles as markers of atherogenicity - all measured in the Brigham Research Assay Laboratory. Visceral fat will be assessed using Dixon MRI technique.

Wellbeing: We will assess mood, anxiety, pain, and life satisfaction as measures of wellbeing. Mood will be assessed using Patient Health Questionnaire (PHQ-9), a 9-item scale that assesses mood and depressive symptoms. We will assess anxiety using GAD-7. Modified Brief Pain Inventory (BPI), a validated measure of pain in SCI, assesses pain intensity (sensory dimension) and interference with function (reactive dimension). Satisfaction with Life Scale is a 5-item scale that assesses happiness with life. Loneliness will be assessed using the Three-Item Loneliness Scale.

Study Population: This proof-of-concept trial will enroll 88 community dwelling men and women with SCI, 19 to 70 years of age, motor C7-T12 cervical and thoracic, AIS A, B, C, or D, 6 months or later after a SCI.

The trial plans to randomize 84 eligible subjects at a single trial site.

Phase: Phase 2

Description of Sites/Facilities Enrolling Participants: This is a single site study that will take place at the Brigham and Women's Hospital in Boston, MA.

Description of Study Intervention: The Home-Based Multimodality Functional Recovery and Metabolic Health Enhancement Program includes training at home consisting of FES-LC plus arm ergometry plus testosterone undecanoate. Testosterone injections will be administered by study staff in the research clinic or by a visiting nurse in the participant's home. The control group will receive FES-LC plus arm ergometry plus placebo injections.

Study Duration: Approximately 54 months

Participant Duration: Approximately 33 weeks (14 weeks for screening, baseline studies, and Day 1, 16 weeks of intervention, and up to 3 weeks of end of study assessments)

ELIGIBILITY:
INCLUSION CRITERIA

1. Men and women, 19 to 70 years
2. Confirmed cervical and thoracic, AIS A-D who are at least 6 months post-injury and who use a wheelchair as their primary mobility mode
3. Medically stable, able to follow directions
4. Able to provide informed consent.
5. For females of reproductive potential who are sexually active: use of highly effective contraception for at least 1 month prior to Day 1 and agreement to use such a method during study participation and for an additional 12 weeks after the end of intervention.

EXCLUSION CRITERIA

1. Upper extremity musculoskeletal conditions (such as advanced rotator cuff pathology or carpal tunnel syndrome) or neurological disorder that in the assessment of the study investigator would prevent the participant from performing the prescribed arm ergometry.
2. Current fractures in the upper and lower extremity
3. In accordance with the Endocrine Society and ISSAM Guidelines25,52, we will exclude individuals with a contraindication for androgen use:

   * History of prostate or breast cancer
   * Prostate nodule or induration on digital rectal examination (DRE)
   * Prostate specific antigen (PSA) > 4 ng/ml or > 3 ng/ml in individuals at high risk of prostate cancer such as African Americans or those with family history of prostate cancer in first degree relatives, unless there has been a negative prostate biopsy within 3 months
   * Hematocrit > 48%
4. Conditions that would render exercise and FES unsafe or unfeasible such as severe autonomic dysreflexia, severe pressure sores, severe spasticity and severe pain.
5. Body mass index (BMI) > 45 kg/m2
6. Renal dysfunction as indicated by GFR of <50 ml/min, estimated by using the Modification of Diet in Kidney Disease (MDRD) Study equation, in accordance with K/DOQI guidelines
7. Use of testosterone or other anabolic therapies, including DHEA and androstenedione, or rhGH in the preceding 6 months
8. Active cancer requiring therapy and which may limit life expectancy to less than 5 years
9. Psychosis, bipolar disorder, or major untreated depression
10. Dementia (Mini-Mental Status Exam [MMSE] <24)
11. Myocardial infarction (MI) or stroke within 3 months of entry
12. Pacemaker
13. ALT and AST > 3 x upper limit of normal
14. Poorly controlled diabetes as indicated by hemoglobin (Hb)-A1c greater than 9.0% or diabetes requiring insulin therapy
15. Blood thinners such as Coumadin, heparin, rivaroxaban (Xarelto), dabigatran (Pradaxa), lovenox (subcutaneous heparin), apixaban (Eliquis) (aspirin, plavix and other anti-platelet agents are allowed)
16. Systolic blood pressure (BP) > 170 or diastolic BP > 100 mm Hg
17. Current grade 2 or greater pressure ulcers at relevant contact sites
18. Pressure sores or open wounds on the areas that restricts their participation
19. Because the safety of testosterone has not been established in pregnancy and lactation, we will exclude pregnant or lactating women and women of childbearing potential who are sexually active but are unwilling or unable to use a reliable form of contraception. We will perform a blood test to exclude pregnancy at the time of enrollment.
20. Participation in a structured exercise program currently or in the past 2 months and unwilling to stop the structured exercise program if ongoing at time of screening. Specifically, participation in a structured exercise program, currently or in the past 2 months, that involves progressive resistance exercise training of moderate to high intensity or regular endurance exercise of moderate to high intensity, and unwillingness to stop the structured exercise program if ongoing at time of screening.
21. Inability or unwillingness to participate in the exercise training or the assessments of muscle performance and physical performance

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2019-08-23 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
peak aerobic capacity achieved during arm ergometry exercise | change from baseline to 16 weeks
  The change in peak aerobic capacity from baseline to 16 weeks will be measured as the VO2 peak measured during cardiopulmonary testing using arm ergometry exercise.

SECONDARY OUTCOMES:
skeletal muscle and fat mass | 16 weeks
  magnetic resonance imaging (MRI) using the Dixon method
whole body and regional soft tissue lean and fat mass | 16 weeks
  Measured using DXA
maximal voluntary strength in upper extremity | 16 weeks
  1-repetition maximum strength in the seated chest press exercise, measured in force units (Newtons)
Muscle endurance in upper extremity | 16 weeks
  muscle endurance in the seated chest press exercise, measured in number of repetitions to failure
Maximal voluntary power in upper extremity | 16 weeks
  muscle power in the seated chest press exercise, measured in Watts.
Safety Assessment | throughout 16 weeks of subjects participation
  Adverse and Serious Adverse Event recording classified using MEDRA and SOC coding
Self-reported function and mobility | 16 weeks
  self-reported function and mobility measured by the Spinal Cord Injury Function Index (SCI-FI). The score range is 13 to 52, with higher scores indicating better function and mobility.
Mood | 16 weeks
  Patient Health Questionnaire (PHQ-9). The score range is 0 to 27. A higher score indicates more severe depression.
Anxiety | 16 weeks
  Generalized Anxiety Disorder 7-item scale (GAD-7). Score range is 0 to 21. A higher score indicates worse anxiety.
Satisfaction with Life | 16 weeks
  Satisfaction with Life Scale (5 item scale). The score range is from 5 to 35. Higher scores indicate more satisfaction with life.
Loneliness | 16 weeks
  Three-Item Loneliness Scale. Score range is 2 to 8, with a score of 2 indicating the least loneliness and 8 the most loneliness
Pain | 16 weeks
  Brief Pain Inventory (BPI). Score range is 0 to 10. Higher scores indicate worse pain.
Peak aerobic capacity during FES-LC exercise alone | change from baseline to 16 weeks
  Change from baseline in peak V02 aerobic capacity achieved during the functional electrical stimulation -leg cycle (FES-LC) exercise alone
Peak aerobic capacity achieved during combined FES-LC and AE exercise | change from baseline to 16 weeks
  The change from baseline in the V02 peak aerobic capacity during the combined functional electrical stimulation- leg cycling (FES-LC) and arm ergometry (AE) exercise
metabolism measures - fasting glucose A1C | 16 weeks
  The percent fasting glucose A1C at final outcome assessment
metabolism measures - lipoprotein particles | 16 weeks
  lipoprotein particles at final outcome assessment, measured as mg/dL
metabolism measures - insulin sensitivity | 16 weeks
  insulin sensitivity at final outcome assessment, measured as Homeostatic Model Assessment - Insulin Resistance Index.
Chronotropic Index | 16 weeks
  The Chronotropic Index is the slope of heart rate (HR) versus whole body oxygen uptake (VO2) measured while subjects are performing a progressive work test using cycle ergometry.

OTHER OUTCOMES:
Change in total trabecular volumetric bone density in the distal tibia | Change from baseline to 16 weeks
  Change from baseline in total, trabecular volumetric bone density measured using HR-pQCT at the distal tibia
Change in total trabecular volumetric bone density in the distal radius | Change from baseline to 16 weeks
  Change from baseline in total, trabecular volumetric bone density measured using HR-pQCT at the distal radius
Change in total cortical volumetric bone density in the distal radius | Change from baseline to 16 weeks
  Change from baseline in total cortical volumetric bone density measured using HR-pQCT at the distal radius
Change in total cortical volumetric bone density in the distal tibia | Change from baseline to 16 weeks
  Change from baseline in total cortical volumetric bone density measured using HR-pQCT at the distal tibia
Change in bone microarchitecture in the distal tibia and radius | Change from baseline to 16 weeks
  Change from baseline in bone microarchitecture measured using HR-pQCT at the distal tibia and radius
Change in estimated bone strength of the distal tibia | Change from baseline to 16 weeks
  Change from baseline in estimated bone strength of the distal tibia, assessed using microfinite element analysis of the HR-pQCT data
Change in estimated bone strength of the distal radius | Change from baseline to 16 weeks
  Change from baseline in estimated bone strength of the distal radius, assessed using microfinite element analysis of the HR-pQCT data
Change in areal bone mineral density of the hip and lumbar spine | Change from baseline to 16 weeks
  Change from baseline in areal bone mineral density of the hip and lumbar spine using dual-energy X-ray absorptiometry (DXA
Change in serum osteocalcin level | Change from baseline to 16 weeks
  Change from baseline in serum osteocalcin level
Change in PINP level | Change from baseline to 16 weeks
  Change from baseline in procollagen type I N-terminal propeptide (PINP) level
Change in CTX level | Change from baseline to 16 weeks
  Change from baseline in C-terminal telopeptide (CTX) level

CONTACTS AND LOCATIONS:
Overall Officials: Shalender Bhasin, MB BS, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Valderrabano RJ, Pencina K, Shang YV, Echevarria E, Dixon R, Ghattas C, Wilson L, Reid KF, Storer T, Garrahan M, Tedtsen T, Zafonte R, Bouxsein M, Bhasin S. Bone microarchitectural alterations associated with spinal cord injury: Relation to sex hormones, metabolic factors, and loading. Bone. 2024 Apr;181:117039. doi: 10.1016/j.bone.2024.117039. Epub 2024 Feb 5. PMID 38325649
- [Derived] Reid KF, Storer TW, Pencina KM, Valderrabano R, Latham NK, Wilson L, Ghattas C, Dixon R, Nunes A, Bajdek N, Huang G, Skeels SE, Lin AP, Merugumala SM, Liao HJ, Bouxsein ML, Zafonte RD, Bhasin S. A multimodality intervention to improve musculoskeletal health, function, metabolism, and well-being in spinal cord injury: study protocol for the FIT-SCI randomized controlled trial. BMC Musculoskelet Disord. 2022 May 25;23(1):493. doi: 10.1186/s12891-022-05441-3. PMID 35614404